CLINICAL TRIAL: NCT01480011
Title: A Pilot Study of Efficacy of Lactobacillus CD2 Lozenges in Preventing High-dose Chemotherapy Induced Oral Mucositis in Patients Undergoing Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr Atul Sharma, Additional Professor Medical Oncology, Principal Investigator, All India Institute of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P1101
Record Dates: First submitted 2011-11-04; First posted 2011-11-28 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Oral Mucositis
Keywords: Lactobacillus CD2 lozenges; high-dose chemotherapy induced; hematopoietic stem cell transplantation
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lactobacillus lozenges (Experimental): The study drug contains not less than 2x109 (2 billion) viable cells of Lactobacillus CD2 as active ingredient
  Interventions: Drug: lactobacillus CD2 lozenges

INTERVENTIONS:
Drug: lactobacillus CD2 lozenges — The study drug contains not less than 2x109 (2 billion) viable cells of Lactobacillus CD2 as active ingredient
  Other Names: CD#2

SUMMARY:
Patients with various malignancies who are taken up for high dose chemotherapy followed by stem cell transplant (blood and marrow transplant) have very high chances of developing severe oral mucositis (between 95-100%). This mucositis not only causes significant morbidity but also hampers quality of life so much so that patients at times feel difficult to continue treatment.

No definite treatment exists for prevention or treatment of oral mucositis in this group of patients. Though one study has suggested that use of IV palifermin (a keratinocyte growth factor) will reduce duration and severity. Palifermin is very expensive and not available in country. Recently the investigators have shown effectiveness of a probiotic Lactobacillus CD 2 in reducing incidence and severity of chemo-radiotherapy induced mucositis in head and neck squamous cell cancer patients. (Published online in European Journal of Cancer: http://dx.doi.org/10.1016/j.ejca.2011.06.010). No significant toxicity has been reported with its use.

Now, the investigators want to study the efficacy of this drug to reduce severity of mucositis in patients undergoing hematopoietic stem cell transplantation. The drug will be supplied by CD Pharma India Private Limited.

The investigators further give undertaking that study will be carried as per good clinical practices (GCP) and declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 10 and 70 years.
2. Karnofsky Performance Score ≥ 70%.
3. Confirmed histological diagnosis of cancer/leukaemia for which haematopoietic stem cell transplantation is an approved modality of therapy.
4. Patients eligible to receive high-dose chemotherapy as part of conditioning regime.
5. Concomitant co morbid condition if present, controlled by medicines.
6. Serum creatinine 1.8mg/dl.
7. Total bilirubin 2mg/dl.
8. Liver enzymes within three times of normal limit.
9. Expected survival > 6 months.

Exclusion Criteria:

1. Pregnant women and lactating mothers.
2. Patients with history of AIDS
3. Patients who have taken any other investigational product in last 4 weeks.
4. Patients having untreated symptomatic dental infection.
5. Patients with WHO Grade 3 or 4 oral Mucositis.
6. Other serious concurrent illness.
7. Inconclusive histological diagnosis.
8. Patients on anticancer antibiotics.
9. Patients with signs and symptoms of systemic infections.
10. Patient's/guardian's refusal to sign informed consent.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
incidence of grade III and grade IV mucositis | Day 24 of stem cell infusion or complete healing of mucositis
  Determine the incidence of grade III and IV mucositis in patients undergoing allogeneic or autologous haematopoietic stem cell transplantation .

SECONDARY OUTCOMES:
grade I and grade II mucositis | Day 24 of stem cell infusion or complete healing of mucositis
  1. Determine the incidence of Grade I and II mucositis in patients undergoing allogenic or autologous haematopoietic stem cell transplantation.
  2. Duration of and time period for healing of chemotherapy induced oral mucositis.
  3. Determine incidence and severity of dysphagia

CONTACTS AND LOCATIONS:
Overall Officials: Atul Sharma, MD,DM, Principal Investigator — Dr BRA Institute Rotary Cancer Hospital ,All India Institute of Medical Sciences,New Delhi ,India.
Locations (1):
- All India institute of Medical sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Result] Sharma A, Rath GK, Chaudhary SP, Thakar A, Mohanti BK, Bahadur S. Lactobacillus brevis CD2 lozenges reduce radiation- and chemotherapy-induced mucositis in patients with head and neck cancer: a randomized double-blind placebo-controlled study. Eur J Cancer. 2012 Apr;48(6):875-81. doi: 10.1016/j.ejca.2011.06.010. Epub 2011 Jul 6. PMID 21741230
- [Derived] Sharma A, Tilak T, Bakhshi S, Raina V, Kumar L, Chaudhary S, Sahoo R, Gupta R, Thulkar S. Lactobacillus brevis CD2 lozenges prevent oral mucositis in patients undergoing high dose chemotherapy followed by haematopoietic stem cell transplantation. ESMO Open. 2017 Feb 13;1(6):e000138. doi: 10.1136/esmoopen-2016-000138. eCollection 2016. PMID 28848667